CLINICAL TRIAL: NCT06535308
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Single and Multiple Dosing, Dose-escalation, Phase 1 Clinical Trial to Evaluate the Safety/Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics, Food Effect, Ethnic Difference of BnH-015B After Oral Administration in Healthy Adult Korean and Caucasian Male Volunteers and in Patients With Moderate Alzheimer's Disease
Brief Title: BnH-015B Clinical Trial in Moderate Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BnH Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24_BnH-015B_P1
Record Dates: First submitted 2024-07-08; First posted 2024-08-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: The study will proceed sequentially from Cohort 1 through 8, and the decision to proceed to the next dosage level will be determined by the Safety Review Committee (SRC) based on the safety and tolerability results of the previous dose stage
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- BnH-015B 5 mg (Experimental): Cohort 1 / Single-dose
  Interventions: Drug: BnH-015B 5 mg
- BnH-015B 10 mg (Experimental): Cohort 2 / Single-dose
  Interventions: Drug: BnH-015B 10 mg
- BnH-015B 20 mg (Experimental): Cohort 3 / Single-dose
  Interventions: Drug: BnH-015B 20 mg
- BnH-015B 40 mg (Dietary impact) (Experimental): Cohort 4 / Single-dose
  Interventions: Drug: BnH-015B 40 mg (Dietary impact)
- BnH-015B 40 mg (Experimental): Cohort 4-1 / Single-dose
  Interventions: Drug: BnH-015B 40 mg
- BnH-015B 80 mg (Experimental): Cohort 5 / Single-dose
  Interventions: Drug: BnH-015B 80 mg
- BnH-015B 160 mg (Experimental): Cohort 6 / Single-dose
  Interventions: Drug: BnH-015B 160 mg
- BnH-015B 40 mg (MAD) (Experimental): Cohort 7 / Multiple-dose
  Interventions: Drug: BnH-015B 40 mg (MAD)
- BnH-015B 80 mg (MAD) (Experimental): Cohort 8 / Multiple-dose
  Interventions: Drug: BnH-015B 80 mg (MAD)
- BnH-015B 40 mg (Part II) (Experimental): Experimental group 1
  Interventions: Drug: BnH-015B 40 mg (Part II)
- BnH-015B 80 mg (Part II) (Experimental): Experimental group 2
  Interventions: Drug: BnH-015B 80 mg (Part II)
- BnH-015B Placebo (Part II) (Placebo Comparator): Placebo group
  Interventions: Drug: BnH-015B Placebo (Part II)

INTERVENTIONS:
Drug: BnH-015B 5 mg — Korean / 3 on BnH-015B, 1 on placebo
  Arms: BnH-015B 5 mg
Drug: BnH-015B 10 mg — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 10 mg
Drug: BnH-015B 20 mg — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 20 mg
Drug: BnH-015B 40 mg (Dietary impact) — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 40 mg (Dietary impact)
Drug: BnH-015B 40 mg — Caucasian / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 40 mg
Drug: BnH-015B 80 mg — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 80 mg
Drug: BnH-015B 160 mg — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 160 mg
Drug: BnH-015B 40 mg (MAD) — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 40 mg (MAD)
Drug: BnH-015B 80 mg (MAD) — Korean / 6 on BnH-015B, 2 on placebo
  Arms: BnH-015B 80 mg (MAD)
Drug: BnH-015B 40 mg (Part II) — Korean / 9 subjects
  Arms: BnH-015B 40 mg (Part II)
Drug: BnH-015B 80 mg (Part II) — Korean / 9 subjects
  Arms: BnH-015B 80 mg (Part II)
Drug: BnH-015B Placebo (Part II) — Korean / 6 subjects
  Arms: BnH-015B Placebo (Part II)

SUMMARY:
BnH-015B is a small molecule compound that targets the GluN2B binding site on NMDA receptors and positively modulates. BnH-015B has shown, through nonclinical trials, to improve symptoms of cognitive decline by regulating the BDNF/TRKβ and microglia-mediated IL-33/OPN signaling pathways; therefore, it is expected to be a promising new drug that can significantly improve symptoms associated with Alzheimer's disease, including memory loss.

DETAILED DESCRIPTION:
Given that existing treatments for Alzheimer's disease only temporarily alleviate symptoms or delay cognitive decline, there is an urgent need for new therapeutic options. Based on the aforementioned safety and efficacy study results, BnH Research Co., Ltd. intends to conduct this phase 1 clinical trial as the first-in-human study of BnH-015B to evaluate its safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* [Part I] Young adults: Healthy Korean or Caucasian male volunteers aged between 19 and 45 at the time of screening
* [Part II] Individuals aged between 55 and 85 years at the time of informed consent
* [Part II] The subject must be diagnosed with probable AD dementia according to the National Institute of Aging and Alzheimer Association (NIA-AA) diagnostic guidelines and must meet all of the following clinical criteria: MMSE score: 10-19, CDR-Global Score: 2
* [Part II] Patients who are positive for P-tau181 and osteopontin in serum at the time of screening and are confirmed as amyloid positive via amyloid PET
* [Part II] Patients diagnosed within the last 5 years prior to screening
* [Part II] The subject (or the subject's legal representative) and caregiver must sign the consent for participation in the study, and the same caregiver must assist the subject throughout the entire study period and be continuously available for contact
* [Part II] Individuals who possess sufficient vision, hearing, language ability, motor function, and comprehension to follow the test procedures in the investigator's judgment
* [Part I&II] Individuals who weigh between 55.0 kg and 90.0 kg and have a body mass index (BMI) of 18.0 kg/m2 to 30.0 kg/m2 at the time of the screening
* [Part I&II] Individuals who have received a full explanation about this clinical trial, completely understand it, and voluntarily decide to participate and agree in writing to follow the instructions (however, for Part II, consent from a guardian can be substituted for this)
* [Part I&II] Individuals deemed suitable as subjects for this study by the investigator based on physical examinations, clinical laboratory tests, and medical history evaluations

Exclusion Criteria:

* [Part II] Patients with a history of unstable angina, myocardial infarction, progressive chronic heart failure (New York Heart Association class III or IV), or clinically significant electrocardiographic abnormalities within the year prior to screening
* [Part II] Patients with a history of vascular dementia
* [Part II] Patients diagnosed with dementia or cognitive impairment not related to Alzheimer's disease, including but not limited to significant head trauma, alcohol abuse, frontotemporal dementia, Huntington's disease, Parkinsonian syndromes (e.g., Parkinson's disease, Lewy body dementia), significant cerebrovascular disease, and/or significant seizure disorders
* [Part II] Patients with psychotic symptoms primarily due to conditions other than Alzheimer's disease causing dementia (e.g., schizophrenia, schizoaffective disorder, delusional disorder, or mood disorders with psychotic symptoms)
* [Part II] Patients who must take contraindicated medications throughout the entire study period
* [Part II] Patients who have used cognitive-impairing, long-term permissible concomitant medications (e.g., antidepressants, anticonvulsants, atypical and typical antipsychotics, benzodiazepines) in unstable doses for at least 8 weeks prior to screening visit and during the screening period
* [Part II] Patients who have been vaccinated (including COVID-19 vaccines and booster shots) within 5 days prior to the administration of the investigational product
* [Part I&II] Individuals with clinically significant diseases or medical history in systems such as hepatobiliary, renal, neurological, immune, respiratory, gastrointestinal, endocrine, hematologic/oncologic, cardiovascular, urogenital, or psychiatric systems (however, elderly individuals aged 65 and over who have mild medical histories may participate if the investigator determines that they can discontinue medication at least 2 weeks or five half-lives prior to the first expected administration date.)
* [Part I&II] Individuals with gastrointestinal diseases (such as Crohn's disease, ulcers, gastritis, gastric spasms, and gastroesophageal reflux disease) or a history of surgery (except for simple appendectomies or hernia surgeries) that may affect the safety/tolerability and pharmacokinetic evaluations of the investigational product
* [Part I&II] Individuals who have hypersensitivity reactions or have a clinically significant history of hypersensitivity reactions to drugs that contain the ingredient of the investigational product (BnH-015B) and those in the same class (NMDAR modulator) and other medications (such as aspirin and antibiotics)
* [Part I&II] Individuals with positive results in serum tests (hepatitis B, hepatitis C, human immunodeficiency virus (HIV), syphilis)
* [Part I&II] Individuals with a history of alcohol or drug abuse, or positive results for abused drugs in a urine drug screening test
* [Part I&II] Individuals who exhibit significant abnormalities in neurological examinations conducted at the time of screening
* [Part I&II] Individuals who show the following vital sign values when measured in a seated position after at least 3 minutes of rest: Systolic blood pressure < 80 mmHg or > 139 mmHg, Diastolic blood pressure < 45 mmHg or > 89 mmHg
* [Part I&II] Individuals who exhibit a QT/QTc interval > 450 msec or clinically significant abnormal rhythm findings on an electrocardiogram during screening
* [Part I&II] Individuals who show one or more of the following results in clinical laboratory tests during screening including additional tests: Blood levels of AST (SGOT), ALT (SGPT) > 1.5 times the upper limit of the normal range, eGFR calculated using the CKD-EPI equation: < 60 mL/min/1.73m2
* [Part I&II] Individuals who have taken any prescription drugs or herbal medicine within 2 weeks prior to the planned administration date of the investigational product, or any over-the-counter (OTC) drugs, dietary supplements including liver function aids, or vitamin preparations within 1 week (however, the investigator may choose to enroll the subject if other conditions are deemed appropriate), or are expected to take such substances
* [Part I&II] Individuals who have taken enzyme-inducing drugs like barbiturates or enzyme-inhibiting drugs like clarithromycin within 1 month prior to the planned administration date of the investigational product
* [Part I&II] Individuals who have participated in another clinical trial (including bioequivalence studies) and received an investigational product within 6 months prior to the planned administration date of the investigational product
* [Part I&II] Individuals who have donated whole blood within 2 months or components of blood within 1 month or received a blood transfusion within 2 months prior to the planned administration date of the investigational product
* [Part I&II] Current smokers (however, those who quit smoking at least 3 months prior to the planned administration date of the investigational product can be enrolled as subjects) or individuals who cannot abstain from smoking during the entire study period
* [Part I&II] Individuals who regularly consume alcohol (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol from 3 days prior to the first expected administration date until the end of the study
* [Part I&II] Individuals who have regularly consumed excessive caffeine (exceeding 5 units/day) or cannot abstain from consuming caffeine-containing foods and beverages (such as coffee, tea (black, green, etc.), carbonated drinks, coffee milk, energy drinks, and sports drinks) from 3 days prior to the planned administration date of the investigational product until the end of the study
* [Part I&II] Individuals who have consumed grapefruit, grapefruit juice, or grapefruit-containing foods from 3 days prior to the planned administration date of the investigational product until the end of the study, or cannot abstain from consuming such grapefruit-containing foods during this period
* [Part I&II] Individuals with unusual dietary habits (e.g., drinking more than 1 liter of grapefruit juice per day) or who cannot consume the standardized diet provided by the clinical trial center during the hospitalization period
* [Part I&II] Individuals who, or whose spouses (or partners), are unable or unwilling to use medically acceptable contraceptive methods during the entire study period and for at least 3 months after the last administration of the investigational product, or do not agree to refrain from donating sperm or eggs (applicable only to Part II) during this period
* [Part I&II] Individuals with dysphagia or who are unable to swallow multiple pills
* [Part I&II] Individuals deemed unsuitable for participation by the investigator for any other reason not specified above

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences, affected participants with adverse events | Through study completion, an average of 14 days
  Safety/tolerability evaluation
Pharmacokinetic (PK) plasma concentration of BnH-015B | 0 hours(pre-dose), 15 minutes, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours post-dose

SECONDARY OUTCOMES:
Changes in serum biomarker concentration | Baseline and 14 days after administration

OTHER OUTCOMES:
Changes in the metabolites of BnH-015B | 0 hours(pre-dose), 15 minutes, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea